CLINICAL TRIAL: NCT06799650
Title: Clinical Study to Evaluate the Efficacy and Safety of Gammora® in Addition to Standard Antiretroviral Treatment for HIV Infection in Antiretroviral Treatment-Naïve Participants
Brief Title: Clinical Trial of Gammora® Plus Antiretroviral Treatment for HIV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Code Pharma (Industry)
Responsible Party: Principal Investigator, Ricardo Sobhie Diaz, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-22-03
Record Dates: First submitted 2024-06-10; First posted 2025-01-29 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-04

CONDITIONS: HIV Seropositivity
Keywords: HIV cure; integrase peptide; proviral HIV DNA; apoptosis; antiretroviral therapy
MeSH Terms: conditions — HIV Seropositivity | interventions — Tenofovir; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gammora® arm (Experimental): 16-mer HIV integrase-derived peptide associated with Tenofovir/3TC + boosted darunavir antiretroviral regimen
  Interventions: Drug: Gammora®
- Control arm (No Intervention): Tenofovir/3TC + boosted darunavir antiretroviral regimen

INTERVENTIONS:
Drug: Gammora® — Gammora® SC + Tenofovir/3TC + darunavir+ritonavir
  Other Names: Tenofovir; 3TC; Darunavir; Ritonavir
  Arms: Gammora® arm

SUMMARY:
The goal of this phase II, open-label, randomized, controlled clinical trial is to evaluate the impact of Gammora®, a 16-mer HIV integrase-derived peptide associated with a boosted darunavir antiretroviral regimen compared Gammora® arm) to a boosted darunavir antiretroviral regimen only (control arm) in the estimated HIV reservoir among antiretroviral naïve people living with HIV. The main questions it aims to answer are:

1. Will the proviral (total) HIV-1 DNA decrease rapidly in the Gammora® arm compared to the control arm?
2. Will the apoptosis markers evaluated in the CD4+ T cell by flow cytometry increase in the Gammora® arm compared to the control arm? Forty antiretroviral naïve viremic people with HIV with CD4+ T cell counts >350 cells/mL will be randomized to receive 20 mg of Gammora® in 2mL SC solution plus Tenofovir/3TC and Darunavir 800mg+Ritonavir 100mg (Gammora® arm) or antiretroviral only (control arm). In the Gammora® arm, participants had a 2-week Gammora® monotherapy lead-in period with Gammora® given daily before antiretroviral treatment is started, followed by 12 weeks of antiretroviral therapy plus Gammora® given every other day. The first two weeks of the trial (lead-in period for the Gammora® arm) were labeled w-2 and w-1 for both groups, and blood samples were collected for both groups. w0 denotes the week ART was started in both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection;
2. Antiretroviral naive;
3. HIV Viral load > 1.000;
4. CD4+ T cell counts >350 cells/mm3;
5. Body weight > 50 Kg;
6. Signed informed consent form.

Exclusion Criteria:

1. BMI < 18.5 kg/m2 at screening;
2. Coinfection with HBV (HBsAg +) or HCV;
3. Any significant acute illness within one week before the first visit.
4. Use of any immunomodulatory therapy (including interferon), systemic steroids, or systemic chemotherapy within four weeks before screening;
5. Active malignancy or malignancy in follow-up.
6. Changes in safety tests: neutrophil count < 1,000 u/L; Hb < 9.0 gm/dl; platelet count < 75,000 u/L; creatinine > 1.5 mg/dl, direct bilirubin > 85 μmol/L, AST or ALT > 2.5 X UNL;
7. Potential allergy or hypersensitivity to the components of the Gammora® formulation.
8. Participation in another clinical trial within 12 months before screening.
9. Any medical condition that makes the participant unsuitable for the study or increases the risk of participation at the investigator's discretion.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Transgender women
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Total Proviral HIV DNA quantitation | Weekly from time of randomization for 27 consecutive weeks
  Total HIV DNA measured by qPCR
Episomal Proviral HIV DNA quantitation | Weekly from time of randomization for 27 consecutive weeks
  Episomal HIV DNA measured by qPCR
Apoptosis markers | Three times per week during from randomization to week 3 and weekly from that point through week 27
  Evaluated by flow cytometry exclusively in the CD4+ T cell gates, using the PE Annexin V Apoptosis Detection kit (BD Biosciences)

SECONDARY OUTCOMES:
HIV Viral load | Weekly from time of randomization for 27 consecutive weeks
  Viral RNA in copies per mL of plasma
CD4 T cell counts | Weekly from time of randomization for 27 consecutive weeks
  CD4+ T cell count per mL
CD8 T cell counts | Weekly from time of randomization for 27 consecutive weeks
  CD8+ T cell count per mL
Levels of Lymphocyte T Cell activation markers (CD38 and HLA-DR in CD4 and CD8+ T cells) for each participant | Weekly for 12 weeks and every 4 weeks after that
  CD38 and HLA-DR in CD4 and CD8+ T cell lymphocytes by flow cytometry
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Weekly for 12 weeks and every 4 weeks after that
  A list of adverse events, separated by treatment-related or not treatment-related as assessed by CTCAE v4.0 per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo S Diaz, M.D., Ph.D., Principal Investigator — Universidade Federal de São Paulo,
Locations (1):
- RDSS, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data to be shared will be anonymized demographic data and outcome measure results.

REFERENCES:
- [Background] Levin A, Hayouka Z, Friedler A, Loyter A. Specific eradication of HIV-1 from infected cultured cells. AIDS Res Ther. 2010 Aug 19;7:31. doi: 10.1186/1742-6405-7-31. PMID 20723214
- [Background] Levin A, Hayouka Z, Helfer M, Brack-Werner R, Friedler A, Loyter A. Peptides derived from HIV-1 integrase that bind Rev stimulate viral genome integration. PLoS One. 2009;4(1):e4155. doi: 10.1371/journal.pone.0004155. Epub 2009 Jan 7. PMID 19127291
- [Background] Levin A, Hayouka Z, Helfer M, Brack-Werner R, Friedler A, Loyter A. Stimulation of the HIV-1 integrase enzymatic activity and cDNA integration by a peptide derived from the integrase protein. Biopolymers. 2010 Aug;93(8):740-51. doi: 10.1002/bip.21469. PMID 20517955
- [Background] Rizza SA, Badley AD. HIV protease inhibitors impact on apoptosis. Med Chem. 2008 Jan;4(1):75-9. doi: 10.2174/157340608783331443. PMID 18220972